CLINICAL TRIAL: NCT01799343
Title: Water Immersion and Changes in the Fetoplacental Circulation. A Case-Control Study With the Case as it's Own Control.
Brief Title: Water Immersion and Changes in the Fetoplacental Circulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Dorthe Thisted, Specialist trainee, Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H-4-2010-139; 2011-41-5889 (Registry Identifier: The Danish Data Protection Agency)
Record Dates: First submitted 2013-02-21; First posted 2013-02-26 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Pregnancy; Immersion
Keywords: Prenatal care; Blood flow velocity; Hydrotherapy; Fetalplacental circulation; Uteroplacental circulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Immersion into water (Experimental): Normal healthy singleton pregnant women. The case serves as its own control. Measurements of mean arterial pressure, deepest vertical pocket of amnion fluid and Doppler flow in the umbilical and uterine arteries will be assessed before immersion (Baseline), during immersion (Immersion) and after immersion (Post-immersion).
  Interventions: Other: Immersion into water

INTERVENTIONS:
Other: Immersion into water — Measurements of mean arterial pressure, deepest vertical pocket of amnion fluid and Doppler flow in the umbilical and uterine arteries will be assessed before immersion, during immersion and after immersion.

SUMMARY:
Pregnant women with pre-eclampsia and growth restricted fetuses often have a reduced function of the placenta. This is accompanied by an increased perinatal mortality and morbidity.

By ultrasound it is possible to measure blood flow and vascular resistance in both the fetal umbilical cord and in the blood vessels supplying the uterus. A high resistance in these vessels occur before the child is severely affected.

By immersion in water extracellular fluid is redistributed back into the circulation, and central blood volume increases. Previous studies have shown that maternal minute-volume increases, while blood pressure drops slightly. Also an increased amniotic fluid has been recorded. This has been interpreted as an expression of increased renal blood flow. Immersion into water could increase blood flow in the vessels supplying the uterus and thus increase blood flow to the child.

The investigators aim to clarify this by examining blood flow and resistance in the blood vessel supplying the uterus and in the umbilical cord, while the participant is immersed into water. Initially, 25 healthy women with an uncomplicated singleton pregnancy recruited from the Department of Obstetrics and Gynaecology: Hvidovre University Hospital, Denmark, will be examined. The participant will act as its own control and measurements above water and immersed will be conducted at the same study session.

Ultimately the investigators seek to contribute to a non-invasive option for prolonging those pregnancies where the fetus and/or maternal condition requires delivery several weeks before term, and where immersion of the pregnant woman in the water a few hours one to several times daily, may prolong the pregnancy the required number of hours/days for antenatal steroid treatment to be sufficient.

There are no risks associated with the study and the project team considers it ethical to implement this. The study is not supported by pharmaceutical companies or other groups with economic interests. The project group itself has taken the initiative to study.

DETAILED DESCRIPTION:
Intrauterine growth retardation and preeclampsia are major causes of neonatal mortality, morbidity and later neurological sequelae. The conditions are associated with an increased resistance to blood flow in the placenta, that can be detected by an increase in pulsatility index (PI) in the umbilical artery (1).

When Doppler flow is assessed in the uterine arteries, increased resistance in the uteroplacental circuit is indicated both by an increase in PI and by a change in the flow velocity waveform, which can be seen as a "notch" in early diastole.

In the 2nd trimester, the invasion of trophoblasts and the remodeling of the uterine spiral arteries are complete. Persistence of a bilateral notch beyond the 24th week of gestation is associated with an increased risk of intrauterine growth retardation and preeclampsia. Even though the risk persists, the notch usually disappears later in pregnancy (2).

When the non-pregnant body is immersed in water, extracellular fluid is redistributed back into the circulation. Central blood volume, cardiac output, renal perfusion and urine output increase and the blood pressure falls (3-7).

The same changes occur in the pregnant women. However the increased diuresis is strongly correlated with the degree of the pregnancy edema, which decreases substantially (8), and the amount of amniotic fluid increases (9). The changes all occur within minutes (8), but are transient and return to conditions before immersion within 1-2 hours after the pregnant woman has come out of the water.

The changes in the above parameters are significant but less pronounced in pregnant women with preeclampsia than in pregnant women without the condition (11). None of the experiments showed changes in the fetal heart rate.

Because of the physiological changes that take place when pregnant women are immersed in water, several authors have speculated whether immersion has a positive effect on the uteroplacental circuit (8,10,12).

There are no published data on Doppler flow measurements in the umbilical artery and the uterine arteries during water immersion.

The aim of the present study is to evaluate the effect of immersion on the fetoplacental and uteroplacental circuits in healthy pregnant women, using Doppler flow measurements in the umbilical artery and uterine arteries.

Materials From the Department of Obstetrics and Gynecology, Hvidovre University Hospital, Denmark, we recruit 25 healthy women with an uncomplicated singleton pregnancy. Gestational age was between 26 and 38 weeks. All participants will have a normal first trimester combined screening and a normal second trimester ultrasound scan for fetal abnormalities. Within the last 2 weeks prior to participation, fetal weight will be estimated, and only woman with fetuses of normal weight (within the 95 percentile) will be included.

Methods The study is performed at the labor ward at Hvidovre Hospital, Denmark. If fetal weight has not been estimated by an ultrasound examination within the last 2 weeks, fetal weight will be estimated on the day of the study. In order to exclude an on-going infection, the temperature is measured and the urine examined in all participants on the day of the study.

The same experienced sonographer performs all examinations, and the same Bruel & Kjaer ultrasound scanner, suitable for scanning under water, is used in all participants.

Each participant has five recordings of blood pressure, pulse, saturation, deepest vertical pocket (DVP) of amniotic fluid and Doppler flow in the umbilical artery and uterine arteries. All recordings are obtained during the same study session. Doppler ultrasound measurements of umbilical and uterine arteries are obtained by pulsed wave ultrasound using an insonating angle as close to 0 degrees as possible. The Doppler measurements on the uterine arteries are obtained approximately one centimeter from the crossing of the iliac arteries. The pulsatility index (PI) is calculated automatically by the machine using the formula (systolic velocity-diastolic velocity)/mean velocity. PI of the uterine artery is calculated as the mean PI of the left and the right uterine artery.

For immersion, a regular bathtub is used. The tub is filled with thermo-neutral tap water (35.0 °C +/- 0.5 °C). The temperature of the water is measured every 10 minutes, and kept thermo-neutral during the period of immersion.

The participants are placed in a supine position outside the bathtub and the first recordings are obtained (T0). Afterwards the participants are immersed in water, placed in a supine position, and measurements are repeated after 5 min (T5) and 25 min (T25) in water. All measurements are repeated with the participant in a supine position outside the bathtub 15 min (T40) and 30 min (T55) after immersion.

All recordings of Doppler flow curves and measurements of amniotic fluid (DVP) are saved on an USB stick. An experienced specialist in fetal medicine, who is not present at the investigation, validates each recording blindly. Any recording not eligible for approval is redefined as a missing value.

Statistical analysis Because the measurements taken before, during and after immersion, are made in the same patient during the same study session, and with the same ultrasound apparatus, each participant act as their own control.

Data are expressed as means +/- standard error of the mean (SEM). The first recording, T0, was defined as baseline. Comparisons between the respective recordings, T0-T55, are done using a two-tailed paired t-test on raw data. P-values < 0.05 are considered significant. For calculation, STATA 12.1 (13) is used.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnant women
* Normal weight fetuses
* Normal first trimester combined screening
* Normal second trimester ultrasound scan for fetal abnormalities

Exclusion Criteria:

* Cardiovascular disease
* Thyroid disease
* Abuse of medication, alcohol- or drugs
* Medical treatment of hypertension
* Medical treatment of depression or any other psychiatric disorder
* Ongoing infection
* Placenta previa
* Cerclage
* Premature rupture of membranes
* Body mass index above 35

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Changes in pulsatility index in umbilical and uterine arteries following immersion into water | After 5 and 25 minutes of immersion and after 15 and 30 past immersion

SECONDARY OUTCOMES:
Changes in maternal mean arterial pressure and in amniotic fluid following immersion into water | After 5 and 25 minutes of immersion and after 15 and 30 minutes past immersion

CONTACTS AND LOCATIONS:
Overall Officials: Niels Jørgen Secher, Prof., MD, Study Chair — Dep. Gynaecology and Obstetrics, Hvidovre University Hospital; Dorthe LA Thisted, MD, Principal Investigator — Dep. Gynaecology and Obstetrics, Hvidovre University Hospital
Locations (1):
- Dep. Gynaecology and Obstetrics, Hvidovre University Hospital, Hvidovre, Hvidovre, Denmark

REFERENCES:
- [Background] Marsal K. Obstetric management of intrauterine growth restriction. Best Pract Res Clin Obstet Gynaecol. 2009 Dec;23(6):857-70. doi: 10.1016/j.bpobgyn.2009.08.011. Epub 2009 Oct 24. PMID 19854682
- [Background] Cnossen JS, Morris RK, ter Riet G, Mol BW, van der Post JA, Coomarasamy A, Zwinderman AH, Robson SC, Bindels PJ, Kleijnen J, Khan KS. Use of uterine artery Doppler ultrasonography to predict pre-eclampsia and intrauterine growth restriction: a systematic review and bivariable meta-analysis. CMAJ. 2008 Mar 11;178(6):701-11. doi: 10.1503/cmaj.070430. PMID 18332385
- [Background] Epstein M, Miller M, Schneider N. Depth of immersion as a determinant of the natriuresis of water immersion. Proc Soc Exp Biol Med. 1974 Jun;146(2):562-6. doi: 10.3181/00379727-146-38147. No abstract available. PMID 4834465
- [Background] Epstein M, Norsk P, Loutzenhiser R, Sonke P. Detailed characterization of a tank used for head-out water immersion in humans. J Appl Physiol (1985). 1987 Aug;63(2):869-71. doi: 10.1152/jappl.1987.63.2.869. PMID 3654446
- [Background] Epstein M, Duncan DC, Fishman LM. Characterization of the natriuresis caused in normal man by immersion in water. Clin Sci. 1972 Aug;43(2):275-87. doi: 10.1042/cs0430275. No abstract available. PMID 5048310
- [Background] Epstein M. Renal, endocrine and hemodynamic effects of water immersion in man. Contrib Nephrol. 1984;41:174-88. doi: 10.1159/000429282. No abstract available. PMID 6570093
- [Background] Greenleaf JE. Physiological responses to prolonged bed rest and fluid immersion in humans. J Appl Physiol Respir Environ Exerc Physiol. 1984 Sep;57(3):619-33. doi: 10.1152/jappl.1984.57.3.619. PMID 6386766
- [Background] Katz VL. Water exercise in pregnancy. Semin Perinatol. 1996 Aug;20(4):285-91. doi: 10.1016/s0146-0005(96)80021-8. PMID 8888454
- [Background] San Juan Dertkigil M, Cecatti JG, Sarno MA, Cavalcante SR, Marussi EF. Variation in the amniotic fluid index following moderate physical activity in water during pregnancy. Acta Obstet Gynecol Scand. 2007;86(5):547-52. doi: 10.1080/00016340601181649. PMID 17464582
- [Background] Kwee A, Graziosi GC, Schagen van Leeuwen JH, van Venrooy FV, Bennink D, Mol BW, Cohlen BJ, Visser GH. The effect of immersion on haemodynamic and fetal measures in uncomplicated pregnancies of nulliparous women. BJOG. 2000 May;107(5):663-8. doi: 10.1111/j.1471-0528.2000.tb13310.x. PMID 10826583
- [Background] Elvan-Taspinar A, Franx A, Delprat CC, Bruinse HW, Koomans HA. Water immersion in preeclampsia. Am J Obstet Gynecol. 2006 Dec;195(6):1590-5. doi: 10.1016/j.ajog.2006.05.007. Epub 2006 Jul 26. PMID 16875643
- [Background] Katz VL. Exercise in water during pregnancy. Clin Obstet Gynecol. 2003 Jun;46(2):432-41. doi: 10.1097/00003081-200306000-00022. No abstract available. PMID 12808393